CLINICAL TRIAL: NCT06471738
Title: Safety and Efficacy of Zanubrutinib in Combination With Rituximab and Venetoclax in Previously Untreated Follicular Lymphoma: An Open Label, Phase 2 Study
Brief Title: Combination of Zanubrutinib, Rituximab and Venetoclax in Patients With Previously Untreated Follicular Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Chief physician., Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-086
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Ann Arbor Stage II Follicular Lymphoma; Grade 1 Follicular Lymphoma; Ann Arbor Stage III Follicular Lymphoma; Ann Arbor Stage IV Follicular Lymphoma; Grade 2 Follicular Lymphoma; Grade 3a Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — zanubrutinib; Rituximab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (zanubrutinib, venetoclax, rituximab) (Experimental): stage I (cycles 1-3, every 4 weeks): zanubrutinib PO 160mg, BID; rituximab IV on day 1.
  stage II (cycles 4-9, every 4 weeks): if complete response : zanubrutinib PO 160mg, BID; rituximab IV on day 1.
  if no complete response : zanubrutinib PO160mg, BID; rituximab IV on day 1 and Venetoclax PO (100mg D1, 200mg D2, and 400mg D3 of cycle 4; 400mg QD).
  Interventions: Drug: Zanubrutinib; Biological: Rituximab; Drug: Venetoclax

INTERVENTIONS:
Drug: Zanubrutinib — BTK inhibitor
Biological: Rituximab — Monoclonal antibody to CD20
Drug: Venetoclax — BCL-2 inhibitor

SUMMARY:
This is a single center, open label, single arm phase II clinical trial. The objective of this study is to assess the feasibility and efficacy of zanubrutinib combined with venetoclax and Rituximab in patients with previously untreated follicular lymphoma (FL) .

DETAILED DESCRIPTION:
Follicular lymphoma (FL)is the most common inert non Hodgkin's lymphoma (iNHL). Their natural courses are slow but highly variable. The standard first-line treatment of advanced FL is based on rituximab. Whether combined with chemotherapy or not, it can induce lasting remission, but it is usually incurable. Although the first-line immunochemotherapy regimen has high efficacy, it also has high toxicity. Cytotoxic chemotherapy is related to many side effects, including bone marrow suppression and immunosuppression, gastrointestinal and cardiac toxicity, neurotoxicity and the occurrence of secondary tumors. About 20% of FL patients relapse within 2 years after first-line chemotherapy. The overall prognosis of these patients is poor. This clinical trial aims to evaluate the feasibility and efficacy of free-chemotherapy regimen (zanubrutinib combined with venetoclax and Rituximab) in patients with previously untreated follicular lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of follicular lymphoma (grades 1, 2, or 3a), untreated
* Stage II, III, or IV disease
* Able and willing to provide written informed consent and to comply with the study protocol
* at least one measurable disease
* Must be in need of therapy as evidenced by at least one of the following criteria:
* Presence of at least one B symptom:

  * Fever (> 38 Celsius [C]) not due to infectious etiology
  * Night sweats
  * Weight loss > 10% in the past 6 months
* Fatigue due to lymphoma
* Splenomegaly (> 13 cm)
* Compression syndrome (ureteral, orbital, gastrointestinal)
* Any of the following cytopenias, due to lymphoma:

  * Hemoglobin ≤ 10 g/dL
  * Platelets ≤ 100 x 10^9/L
  * Absolute neutrophil count (ANC) < 1.5 x 10^9/L
* Pleural or peritoneal effusion
* Lactate dehydrogenase (LDH) > upper limit of normal (ULN) or beta (B)2 microglobulin > ULN
* Other lymphoma-mediated symptoms as determined by the treating physician

Exclusion Criteria:

* ECOG≤ 2
* Absolute neutrophil count (ANC) > 1.0 x 10^9/L
* Platelet count > 50 x 10^9/L
* Prothrombin time (PT)/international normal ratio (INR) < 1.5 x (upper limit of normal) ULN and partial thromboplastin time (PTT) (activated partial thromboplastin time [aPTT]) < 1.5 x ULN (unless abnormalities are unrelated to coagulopathy or bleeding disorder). When treated with warfarin or other vitamin K antagonists, then INR ≤ 3.0)
* Serum aspartate transaminase (AST) and alanine transaminase (ALT) < 3 x upper limit of normal (ULN)
* Creatinine clearance > 30 ml/min calculated by modified Cockcroft-Gault formula
* Bilirubin < 1.5 x ULN unless bilirubin is due to Gilbert's syndrome, documented liver involvement with lymphoma, or of non-hepatic origin, in which case bilirubin should not exceed 3 g/dL
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [B-hCG]) pregnancy test at screening. Women who are pregnant or breastfeeding are ineligible for this study

Exclusion Criteria:

* Known active central nervous system lymphoma or leptomeningeal disease
* Follicular lymphoma with evidence of diffuse large B-cell transformation
* Grade 3b follicular lymphoma
* Any prior history of other malignancy besides follicular lymphoma
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* Patients who have undergone major surgery within 14 days
* The researchers believe that it is not advisable for the participant to take part in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
CR rate | Within 6 months of therapy completion
  Determined by PET/CT based on Cheson, Lugano classification 2014 as assessed by the investigator. The number and percentage of subjects with a CR will be tabulated.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Within 6 months of therapy completion
  CR + partial response (PR), determined by PET/CT based on Cheson, Lugano classification 2014 as assessed by the investigator. The number and percentage of subjects with an ORR will be tabulated.
Progression-free survival | up to two years
  PFS is defined as the duration from date of treatment initiation to date of disease progression or death from any cause
Overall survival | up to two years
  PFS is defined as the duration from date of treatment initiation to date of death from any cause
Incidence of Treatment-Emergent Adverse Events | Up to 90 days after the last dose of study drugs
  Incidence of subjects occuring treatment related adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department and Hematology Department of Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No